CLINICAL TRIAL: NCT01258166
Title: Traumatic Ulnar Translocation of the Carpus: Early Diagnosis and Treatment
Brief Title: Traumatic Ulnar Translocation of the Carpus
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, John Berschback, Resident Physician, Northwestern University
Other Study IDs: STU00023348
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Traumatic Ulnar Translocation of the Carpus
MeSH Terms: interventions — Surgical Procedures, Operative; Immobilization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Tramuatic ulnar translocation: Patients who suffered a traumatic ulnar translocation following injury.
  Interventions: Procedure: Surgery or immobilization

INTERVENTIONS:
Procedure: Surgery or immobilization

SUMMARY:
Ulnar translocation of the carpus is a form of wrist instability where the small bones of the wrist shift out of position. It is well recognized in patients with rheumatoid arthritis, but can also occur after a traumatic event, such as a violent football tackle or a fall from a height. The treatment options vary considerably, and there is no consensus of how to best address this injury pattern.

Because traumatic ulnar translocation is relatively rare, the diagnosis may be missed or delayed, causing problems for the patient such as persistent pain and loss of function. The investigators present 11 cases of this injury, discuss how to recognize it, and report our results after different treatment methods.

DETAILED DESCRIPTION:
Ulnar translocation of the carpus is a form of wrist instability where the entire carpus translates medially along the inclined plane of the distal radius. This pattern of instability has been well recognized in patients with rheumatoid arthritis as a result of articular erosions and attenuation of wrist ligaments. In contrast, ulnar translocation of the carpus following trauma is seemingly rare, with published accounts limited to case reports and small case series.

The radiographic features of traumatic ulnocarpal translocation have been described and the instability pattern has been reproduced in cadaveric models. However, the recognition of radiocarpal malalignment may be unintentionally missed or delayed owing due to the uncommon nature of the this injury. The investigators present 11 cases of posttraumatic ulnar translocation of the carpus and review criteria for early recognition of the injury and the results following varying treatment methods.

ELIGIBILITY:
Inclusion Criteria:

Patient who suffered traumatic ulnar translocation of the carpus Willing to sign the consent

Exclusion Criteria:

Patients with collagen vascular disease

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who suffered traumatic ulnar translocation of the carpus
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2005-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chicago Center for Surgery of the Hand, Chicago, Illinois, United States

REFERENCES:
- [Background] Rayhack JM, Linscheid RL, Dobyns JH, Smith JH. Posttraumatic ulnar translation of the carpus. J Hand Surg Am. 1987 Mar;12(2):180-9. doi: 10.1016/s0363-5023(87)80268-x. PMID 3559067
- [Background] Wollstein R, Wei C, Bilonick RA, Gilula LA. The radiographic measurement of ulnar translation. J Hand Surg Eur Vol. 2009 Jun;34(3):384-7. doi: 10.1177/1753193408101465. Epub 2009 Mar 25. PMID 19321529
- [Background] Yang Z, Mann FA, Gilula LA, Haerr C, Larsen CF. Scaphopisocapitate alignment: criterion to establish a neutral lateral view of the wrist. Radiology. 1997 Dec;205(3):865-9. doi: 10.1148/radiology.205.3.9393549.
- [Background] Bellinghausen HW, Gilula LA, Young LV, Weeks PM. Post-traumatic palmar carpal subluxation. Report of two cases. J Bone Joint Surg Am. 1983 Sep;65(7):998-1006. PMID 6885879
- [Background] Mulier T, Reynders P, Broos P, Fabry G. Posttraumatic ulnar translation of the carpus. A case report. Acta Orthop Scand. 1992 Feb;63(1):102-3. doi: 10.3109/17453679209154862. PMID 1738960
- [Result] McMurtry RY, Youm Y, Flatt AE, Gillespie TE. Kinematics of the wrist. II. Clinical applications. J Bone Joint Surg Am. 1978 Oct;60(7):955-61. PMID 701344